CLINICAL TRIAL: NCT04254705
Title: Response to CFTR-modulators in Intestinal Organoids of Patients With CF Having at Least One R334W Mutation
Brief Title: Organoid Study R334W
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes in modulator landscape
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry); KU Leuven (Other); University of Lisbon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ORGANOID-R334W
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2020-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: For stratification of subjects in the subsequent clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Subjects with CF and R334W mutation (Other): Subjects with CF and R334W mutation
  Interventions: Procedure: Rectal Biopsy

INTERVENTIONS:
Procedure: Rectal Biopsy — Suction biopsy or forceps biopsy

SUMMARY:
In contrary to what is seen in FRT cells, rectal organoids of patients with a R334W mutation do respond to CFTR modulators ivacaftor and lumacaftor. The present study will investigate the response to modulators in organoids of 30 patients with CF and a R334W mutation, to allow further stratificaton for a future clinical trial assessing the clinical effect of ivacaftor/tezacaftor in patients with CF and a R334W mutation.

DETAILED DESCRIPTION:
Rationale: CF is caused by mutations in the 'Cystic Fibrosis Transmembrane Conductance Regulator (CFTR)' channel that codes for the CFTR protein, an anion channel. More than 2000 different CFTR mutations have been described. CFTR modulator drugs treat the underlying protein defect by improving folding and trafficking of nascent protein (corrector) or by improving channel opening at the cell membrane (potentiator). In the European Union, treatment with CFTR modulators has only been approved for patients who are homozygous for F508del or carry a mutation of class III or one of a limited number of residual function mutations.

The R334W-CFTR mutation is a rare mutation (270 subjects in the European CF Registry ECFSPR), described in CFTR2 as disease causing. Clinically there is evidence for residual CFTR function in these subjects since only 36% of the patients with R334W are pancreatic insufficient and the mean age of all patients in the CFTR2 database is a bit older (22 years) than patients with CF and 2 known disease causing mutations (20 years). On the other hand, patients with R334W have on average a high sweat chloride (mean 95 mmol/L) and severe lung disease; their mean FEV1 reported to the CFTR database [1] is very similar to that of other patients with the F508del CF causing mutation. In the Leuven clinic we have one subject with R334W/F508del who is 60 year old and has very severe lung disease (FEV1 in the low 40s).

When studied in FRT (Fisher rat thyroid) cells and compared to wild type, the R334W mutation is reported to give rise to normal levels of protein at the cell membrane, but very much decreased function (short circuit current measurement) of 1.3% of wild type. On the other hand there is very limited rescue of CFTR function after addition of the potentiator ivacaftor: from 1% to 5 % of normal.

In contrast with expression in heterologous systems, intestinal organoids allow study of CFTR function in patient specific material. When tested in intestinal organoids from the patient with F508del/R334W in the Leuven clinic, this mutation resulted in some residual function documented by forskolin induced swelling at higher forskolin concentrations, even before addition of CFTR potentiator or corrector. However, addition of ivacaftor and to a lesser degree lumacaftor results in moderate to good rescue of function; the degree of rescue (FIS result) is intermediate between that seen in F508del homozygous subjects and class III mutation subjects. Comparable results are obtained in prof M Amaral's lab in 3 subjects compound heterozygous for F508del/R334W (results in nasal cells, and intestinal organoids). A CFTR functional rescue in organoids from a subject with the R334W/R746X is also reported by the Dutch Utrecht group in organoids; the forskolin induced swelling induced by luma/iva was again between the response seen with iva in organoids from subjects with gating mutations and by luma/iva in organoids derived from F508del homozygous subjects. These findings suggest that R334W might be a suitable candidate for TEZ/IVA treatment.

The study described in this protocol will be the first step of a larger project that also includes a clinical trial. With the present study, the response of organoids of patients with mutation R334W to available

CFTR-modulators will be tested to identify the in vitro response. An interventional clinical trial, submitted as a separate protocol, will subsequently assess the response to modulators in vivo in the same patients. The clinical trial is thus not part of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, a subject must meet all of the following criteria:

  1. Male or female with confirmed diagnosis of CF. The subject must have the following:

     a. One or more characteristic phenotypic features, such as chronic cough and sputum production, persistent chest radiograph abnormalities, or airway obstruction manifested by wheezing and air trapping; or a history of CF in a sibling; or a positive newborn screening test result;
  2. Two CFTR mutations identified of which one is R334W OR only the R334W mutation identified and a sweat chloride value above 60 mmol/L
  3. Age 12 years and older
  4. Subject will sign and date an informed consent form (ICF) and or assent (for subjects 12 to 16 years old).

Exclusion Criteria:

* A potential subject who meets any of the following criteria will be excluded from participation:

  1. Subject has one of the following CFTR-mutations:

     G551D, G1244E, G1349D, G178R, G551S, S1251N, S1255P, S549N, S549R, R117H, P67L, R117C, L206W, R352Q, A455E, D579G, 711+3A>G, S945L, S977F, R1070W, D1152H, 2789+5G>A, 3272 26A>G, 3849+10kbC>T
  2. A history of hemorrhoids and recent rectal bleeding
  3. FEV1 above 90% predicted or below 30% predicted during stable disease
  4. History of lung transplantation.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Response to CFTR-modulator in Intestinal Organoids: Increase in Forskolin induced swelling by addition of tezacaftor+ivacaftor after stimulation with Forskolin (0.8 µmol/L) | At study completion (when rectal biopsy is performed or when organoids are retrieved from the biobank and FIS has been performed), an average of 2 months
  Response to tezacaftor+ivacaftor in the Forskolin Induced Swelling (FIS) assay in rectal organoids

CONTACTS AND LOCATIONS:
Overall Officials: François Vermeulen, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (12):
- University Hospital of Leuven, Leuven, Belgium
- France (4):
  - Centre Hospitalier Lyon Sud, Lyon
  - Centre Hospitalier Régional Universitaire Montpellier, Montpellier
  - Hôpital Cochin, Paris
  - Hôpital Necker, Paris
- Italy (5):
  - Instituto G. Gaslini, Genova
  - Fondazione Ospedale Maggiore Policlinico, Milan
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Sapienza university - Centra Fibrosi Cistica Regione Lazio, Roma
  - Azieda Ospedaliera Universitaria Integrata, Verona
- Hospital Santa Maria, Lisbon, Portugal
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No